CLINICAL TRIAL: NCT02880904
Title: Development of a Vulvar Scarring Grading Scale for Lichen Sclerosus
Brief Title: Vulvar Scarring Grading Scale for Lichen Sclerosus
Status: Terminated | Type: Observational
Why Stopped: Investigator is no longer at Northwestern University
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Research Assistant Professor of Dermatology, Northwestern University
Other Study IDs: STU00202270
Record Dates: First submitted 2016-05-04; First posted 2016-08-26 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Lichen Sclerosus; Lichen Sclerosus et Atrophicus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Photography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Photography — Photos will be taken of the vulvar lichen sclerosus lesions.

SUMMARY:
The study aims to validate a vulvar scarring grading scale for lichen sclerosus (LS).

DETAILED DESCRIPTION:
Utilizing the vulvar disorders registry, protocol #STU00001056, the research team seeks to analyze the medical record data, including standard of care vulvar photographs, of the vulvar LS population at Northwestern Memorial Hospital (NMH) and the outpatient clinics of Northwestern Medicine (NM). These photographs will be used to develop a vulvar scarring grading scale for LS. The objective measurement of scarring severity in LS deidentified standard-of-care patient photographs will be correlated with clinical examination findings to assess validity of the grading scale. The development of an objective and standardized grading scale will assist with the longitudinal evaluation of individual disease, assessment of impact of therapy on scarring, and inform treatment modifications. Further, objective grading of scarring would also provide the opportunity to search for potential correlation between QoL scores and severity of clinical states in scarring dermatoses.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at Northwestern Medicine Department of Dermatology and/or Department of Obstetrics and Gynecology, who were seen by Dr. Bethanee Schlosser, and/or other members of the Vulvar Mucosal Specialty Clinic team in any of their respective clinic settings and underwent complete mucocutaneous examination.
* Patients with histologically confirmed vulvar LS.

Exclusion Criteria:

* Patients who refuse complete mucocutaneous examination.
* Patients who refuse recommended diagnostic procedures.
* Pregnant women or prisoners.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects from the Northwestern University Vulvar Mucosal Specialty Clinic, with histologically confirmed diagnosis of vulvar lichen sclerosus
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Scarring severity grading scale for vulvar lichen sclerosus | one year

SECONDARY OUTCOMES:
Correlation of severity of vulvar LS scarring, as documented at time of clinical examination and compared to scores on the LS grading scale, with the patient quality of life at the time of examination. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bethanee J Schlosser, MD, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hansen A, Carr K, Jensen JT. Characteristics and initial diagnoses in women presenting to a referral center for vulvovaginal disorders in 1996-2000. J Reprod Med. 2002 Oct;47(10):854-60. PMID 12418071
- [Result] Gokdemir G, Baksu B, Baksu A, Davas I, Koslu A. Features of patients with vulvar dermatoses in dermatologic and gynecologic practice in Turkey: is there a need for an interdisciplinary approach? J Obstet Gynaecol Res. 2005 Oct;31(5):427-31. doi: 10.1111/j.1447-0756.2005.00314.x. PMID 16176512
- [Result] McPherson T, Cooper S. Vulval lichen sclerosus and lichen planus. Dermatol Ther. 2010 Sep-Oct;23(5):523-32. doi: 10.1111/j.1529-8019.2010.01355.x. PMID 20868406
- [Result] Goldstein AT, Marinoff SC, Christopher K, Srodon M. Prevalence of vulvar lichen sclerosus in a general gynecology practice. J Reprod Med. 2005 Jul;50(7):477-80. PMID 16130842
- [Result] Schlosser BJ, Mirowski GW. Lichen sclerosus and lichen planus in women and girls. Clin Obstet Gynecol. 2015 Mar;58(1):125-42. doi: 10.1097/GRF.0000000000000090. PMID 25608255
- [Result] Bradford J, Fischer G. Long-term management of vulval lichen sclerosus in adult women. Aust N Z J Obstet Gynaecol. 2010 Apr;50(2):148-52. doi: 10.1111/j.1479-828X.2010.01142.x. PMID 20522071